CLINICAL TRIAL: NCT07233408
Title: Tailoring an Online Platform to Promote Evidence-Based Care for Adults With Neurofibromatosis 1 and Low Health Literacy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Principal Investigator, Vanessa Merker, PhD, Assistant Professor of Neurology, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2024P002819; HT9425-23-1-0457 (Other Grant/Funding Number: U.S. Department of Defense)
Record Dates: First submitted 2025-11-14; First posted 2025-11-18 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Neurofibromatosis 1
Keywords: Neurofibromatosis; NF1; Guideline; Primary Care; Annual Care; Low Health Literacy; Healthcare; PCP
MeSH Terms: conditions — Neurofibromatosis 1; Neurofibromatoses

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NF1 Educational Videos (Experimental)
  Interventions: Other: NF1 Educational Videos; Other: Letters about NF1 Care
- Peer Navigator (Experimental)
  Interventions: Other: Peer Navigator; Other: Letters about NF1 Care

INTERVENTIONS:
Other: NF1 Educational Videos — Participants will receive access to NF1 educational videos that further explain NF1 health surveillance recommendations in advance of the patient's annual wellness visit.
  Arms: NF1 Educational Videos
Other: Peer Navigator — Participants will receive a phone or video call from an NF1 peer navigator. The navigator will explain NF1 health surveillance recommendations and coach individuals on how to discuss these recommendations with their provider.
  Arms: Peer Navigator
Other: Letters about NF1 Care — Participants will receive two letters about NF1 care, one for themselves and one for their primary care clinician, to read in advance of the patient's annual wellness visit.

SUMMARY:
This decentralized, randomized study seeks to assess the feasibility, acceptability, and preliminary effectiveness of two approaches to assisting Neurofibromatosis 1 (NF1) patients with low health literacy improve their understanding of NF1 symptoms and care recommendations. Participants will be provided with personalized NF1 care letters for themselves and their doctors, along with either NF1 educational videos or a call with an NF1 peer navigator.

Adults with NF1 from across the U.S. who have upcoming annual wellness visits scheduled with a primary care provider (PCP) are eligible to enroll in the study. To see if you might be eligible, fill out a prescreening survey here: https://redcap.link/nfpeer

DETAILED DESCRIPTION:
Background: Previous studies indicate that patient understanding of NF1 symptoms and screening for health issues such as hypertension, scoliosis, and cancers could be improved. Many individuals with NF1 have learning challenges, complicating their ability to access NF1 information. To address this gap, researchers are evaluating two interventions to promote understanding of NF1 care within adults with low health literacy.

Methods: Enrolled participants will complete baseline survey assessments online before their PCP visit and then be randomized to either the educational videos or peer navigator intervention group. Both groups will be given personalized letters, one for themselves and one for their clinician, that describe NF1 care recommendations. After attending their annual wellness visit, all participants will be asked to complete an online follow-up survey. A small subsample of participants will also be asked to do a virtual qualitative interview. No visits to Massachusetts General Hospital are required for this study.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Currently lives in the United States
* Has a clinical diagnosis of Neurofibromatosis 1
* Speaks English
* Has low health literacy as ascertained by standardized instruments
* Has an in-person, well-person visit (e.g. not a visit to address an acute medical issue) with their primary care provider (PCP) scheduled within the 3 months following their consent

Exclusion Criteria:

* Unwilling or unable to give informed consent
* Is too cognitively impaired to participate in the opinion of the study investigator (e.g. any cognitive or developmental delay that prevents completion of study questionnaires)
* Was enrolled in or is the parent or guardian of a participant enrolled in randomized clinical trial NCT06262113

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-05-30 (Estimated); Study Completion 2026-05-30 (Estimated)

PRIMARY OUTCOMES:
Feasibility of Videos and NF1 Peer Navigator Use as an Addition to My NF Guide | 2 weeks after PCP visit
  * Recruitment (% of people that complete prescreening who are eligible)
  * Willingness to Enroll (% of prescreening-eligible people who enroll)
  * Retention (% of consented individuals who complete both the baseline survey and follow-up survey)
  * Intervention Completion (% of people who watch all videos or complete peer navigator meeting, as applicable based on intervention assigned)

SECONDARY OUTCOMES:
Client Satisfaction Questionnaire (CSQ-8) | 2 weeks after PCP visit
  The CSQ-8 will be used to assess client satisfaction with the My NF Guide/PEER Resource package (i.e. personalized letters and either NF1 educational videos or peer navigator). It consists of 8 items rated on a 4-point Likert scale, yielding scores that range from 8 to 32. Higher scores indicate greater satisfaction with the services provided.
Telehealth Usability Questionnaire (TUQ) | 2 weeks after PCP visit
  The TUQ will be used to evaluate the ease of use, usefulness, and reliability with the My NF Guide/PEER Resource package (i.e. personalized letters and either NF1 educational videos or peer navigator). It consists of 21 items rated on a seven-point Likert scale ranging from "strongly disagree" to "strongly agree," with a higher average score indicating better usability. The overall usability score will be calculated as the mean of all applicable responses, and sub-scores for specific domains such as usefulness, ease of use, and reliability will be computed for detailed analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Vanessa Merker, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Merker VL, Knight P, Radtke HB, Yohay K, Ullrich NJ, Plotkin SR, Jordan JT. Awareness and agreement with neurofibromatosis care guidelines among U.S. neurofibromatosis specialists. Orphanet J Rare Dis. 2022 Feb 10;17(1):44. doi: 10.1186/s13023-022-02196-x. PMID 35144646
- [Background] Merker VL, McDannold S, Riklin E, Talaei-Khoei M, Sheridan MR, Jordan JT, Plotkin SR, Vranceanu AM. Health literacy assessment in adults with neurofibromatosis: electronic and short-form measurement using FCCHL and Health LiTT. J Neurooncol. 2018 Jan;136(2):335-342. doi: 10.1007/s11060-017-2657-8. Epub 2017 Nov 8. PMID 29119424